CLINICAL TRIAL: NCT02146833
Title: A Phase-2, Open-Label Study of Oral Selinexor (KPT-330) in Patients With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: SHIP (Selinexor in Hormone Insensitive Prostate Cancer)
Acronym: SHIP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to enrollment challenges. The termination is not a consequence of any safety concern.
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCP-330-007
Record Dates: First submitted 2014-05-13; First posted 2014-05-26 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer
Keywords: castrate-resistant prostate cancer; prostate cancer; Karyopharm; KPT-330; selinexor
MeSH Terms: conditions — Prostatic Neoplasms | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Selinexor Dosing Regimen 1 (Experimental): 80 mg twice weekly for 4 weeks (8 doses per 28-day cycle)
  Interventions: Drug: Selinexor
- Selinexor Dosing Regimen 2 (Experimental): 80 mg once weekly for 4 weeks (4 doses per 28-day cycle)
  Interventions: Drug: Selinexor
- Selinexor Dosing Regimen 3 (Experimental): 60 mg twice weekly for 2 weeks, then 1 week off (4 doses per 21-day cycle)
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — Comparison of different dosages and dosing schedules of drug.
  Other Names: KPT-330

SUMMARY:
This is an open-label, Phase 2 clinical study of the oral Selective Inhibitor of Nuclear Export (SINE) selinexor (KPT-330) in patients with metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This is a Phase 2, open-label study to explore the effect of selinexor (KPT-330) therapy in patients with metastatic castration-resistant prostate cancer (mCRPC). Approximately 50 patients are planned for enrollment. Patients will receive an oral dose of selinexor on one of three dosing schedules.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the prostate with evidence for skeletal metastases on bone scan and/or CT scan.
* Must have received at least one agent known to impact survival (abiraterone, enzalutamide, etc.).
* Eastern Cooperative Oncology Group (ECOG) less than or equal to (≤ 2) or a Karnofsky Performance Status (KPS) ≥ 60%.
* Serum testosterone levels less than (<) 50 ng/ml.
* Ongoing gonadal androgen deprivation therapy with luteinising hormone-releasing hormone (LHRH) analogues or orchiectomy. Participants, who have not had an orchiectomy, must be maintained on standard dosing of LHRH analogue therapy at appropriate frequency for the duration of the study.
* Progression of disease despite androgen ablation shown by objective, documented evidence of disease progression (excluding prostate-specific antigen [PSA]), defined as one or both of the following:

  1. Soft tissue disease progression defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
  2. Bone disease progression defined by modified Prostate Cancer Clinical Trials Working Group 2 (PCWG2) with two or more new lesions or bone scan
* Discontinuation of all glucocorticoids prescribed to specifically treat prostate cancer (e.g., as a secondary hormonal manipulation) greater than (>) 4 weeks prior to receiving first dose of study drug. Glucocorticoids prescribed for a chronic non-cancer-related illness (e.g., asthma or chronic obstructive pulmonary disease [COPD]) that is well controlled with medical management are permissible to an equivalent of ≤ 10 milligrams (mg) prednisone daily.
* Laboratory requirements:

  1. White blood cell (WBC) count > 3,000/microliter (μL)
  2. Absolute neutrophil count (ANC) > 1,500/μL
  3. Hemoglobin ≥8.0 gram per deciliter (g/dL)
  4. Platelet count ≥150,000/μL
  5. Serum albumin ≥3.0 g/dL
  6. Calculated or measured creatinine clearance > 30 milliliter per minute (mL/min)
* A biopsy documenting prostate cancer in a target lesion (e.g., lymph node, bone lesion, or soft tissue lesion) within 3 months prior to study entry.
* No evidence of chronic or acute disseminated intravascular coagulation or bleeding tendency.
* Participant must be willing and able to comply with protocol requirements. All participants must sign an informed consent indicating that they are aware of the investigational nature of this study.
* Participant must be willing and able to sign an authorization for the release of their protected health information for study purposes.

Exclusion Criteria:

* Histologic variants other than adenocarcinoma in the primary tumor.
* Participants who require or may be expected to require urgent treatment with docetaxel during the study (e.g., participants with visceral metastases).
* Abnormal hepatic function:

  1. Bilirubin > 2 times the upper limit of normal (2 x ULN) (except participants with Gilbert's syndrome [hereditary indirect hyperbilirubinemia] who must not have a total bilirubin of > 3 x ULN)
  2. Aspartate transaminase (AST) and alanine transaminase (ALT) > 2.5 x ULN (except participants with known liver involvement of their mCRPC who must not have an AST and ALT > 5 x ULN)
* Therapy with other hormonal therapy, including any herbal product known to decrease PSA levels (e.g., Saw Palmetto and PC-SPES) within 4 weeks prior to receiving first dose of study drug.
* Therapy with samarium-153, strontium-89, or radium-223 within 8 weeks prior to first dose of study drug.
* Uncontrolled infection or concomitant illness that is not controlled with medical management.
* Prior external beam radiation therapy completed < 3 weeks or single fraction of palliative radiotherapy within 14 days prior to first dose of study drug.
* Any "currently active" second malignancy, other than non-melanoma skin cancer. Participants are not considered to have a "currently active" malignancy, if they have completed therapy and are considered by their physician to be at least less than 30% risk of relapse over next 3 months.
* Active psychiatric illnesses/social situations that would limit compliance with protocol requirements.
* Active or uncontrolled autoimmune disease that may require corticosteroid therapy during study.
* Severely compromised immunological state, including known human immunodeficiency virus (HIV).
* Known acute or chronic hepatitis B or C.
* Chemotherapy and other investigational therapies (targeted or immunotherapy) will require a 3-week washout period before treatment initiation.
* Initiation of bisphosphonate therapy within 4 weeks prior to first dose of study treatment. Participants receiving ongoing bisphosphonate or denosumab therapy must have been on stable doses for at least 4 weeks prior to receiving first dose of study treatment. Participants on stable doses of bisphosphonates who show subsequent tumor progression may continue on this medication.
* Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

  1. History or presence of serious uncontrolled ventricular arrhythmias or presence of uncontrolled atrial fibrillation.
  2. Clinically significant resting bradycardia (< 50 beats per minute).
  3. Any of the following within 3 months prior to study entry: myocardial infarction severe/unstable angina, Coronary Artery Bypass Graft, Grade 3 or 4 Congestive Heart Failure, Cerebrovascular Accident, Transient Ischemic Attack, or Pulmonary Embolism.
  4. Uncontrolled hypertension, as defined by a systolic blood pressure > 160 mm Hg and/or a diastolic blood pressure > 90 mm Hg with or without anti-hypertensive medication.
  5. Previous pericarditis; clinically significant pleural effusion in the previous 12 months or current ascites requiring 2 or more interventions per month.
  6. Angina at rest.
* Any acute toxicities due to prior chemotherapy and/or radiotherapy that have not resolved to a National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE), version 4.03 Grade of ≤ 1. Chemotherapy induced alopecia or Grade 2 neuropathy is allowed.
* Any condition or situation, which in the Investigator's opinion, may put the participant at significant risk, confound the study results, or interfere significantly with the participant's participation in the study.
* Men with a female partner of child-bearing potential, (defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 12 consecutive months), who as a couple are unable or unwilling to employ two forms of highly effective contraception (e.g., male condom with spermicide, diaphragm with spermicide, intra-uterine device). Two methods of contraception must be used by participants and their partners through the study and for 3 months after the end of study treatment.
* Body mass index (BMI) < 1.2 m^2, in order to prevent a participant from receiving a dose of selinexor > 70 mg/m^2.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at single center in United States of America from May 2014 to 01 April 2016. Due to early termination of study, participants in Arm 2 and 3 were not enrolled.
Pre-assignment Details: A total of 20 participants were enrolled and treated in the study, of which 9 participants completed the study.
Groups:
- Arm 1: Selinexor: Participants received a dose of 80 milligrams (mg) selinexor twice weekly orally on Days 1, 3, 8, 10, 15, 17, 22, and 24 of 28-day cycle until study discontinuation due to any reason.
Period: Overall Study
Arm/Group | Arm 1: Selinexor
Started | 20
Completed | 9
Not Completed | 11
Not completed — Death | 10
Not completed — No longer consented to study treatment | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any amount of study drug.
Groups:
- Arm 1: Selinexor: Participants received a dose of 80 mg selinexor twice weekly orally on Days 1, 3, 8, 10, 15, 17, 22, and 24 of 28-day cycle until study discontinuation due to any reason.
Arm/Group | Arm 1: Selinexor
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 17
  Race: Black or African American | 1
  Race: Asian | 1
  Race: Native Hawaiian or Pacific Islander | 0
  Race: American Indian or Alaska Native | 0
  Race: Other | 1
  Race: Unknown | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Clinical Benefit Response (CBR)
Description: CBR was defined as the point estimate of the percentage of participants who had complete response (CR), partial response (PR), or stable disease (SD) at 12 weeks as per the Response Evaluation Criteria in Solid Tumors (RECIST v.1.1; soft tissue lesions). CR: Disappearance of all target lesions. PR: At least a 30 percent (%) decrease in the sum of diameters of target lesions, taken as reference the baseline sum diameter. SD: steady state of disease; non-CR or non-PR or non-progressive disease.
Time Frame: At 12 weeks
Population: Modified intent-to-treat (mITT) population:Participants who received at least 1 dose of study drug and had at least 1 post-baseline efficacy assessment. Participants who received at least 1 dose of study drug, but discontinued treatment prior to first efficacy follow-up assessment due to death, toxicity, or disease progression were also included.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: Selinexor
Number analyzed (Participants) | 20
Percentage of participants | 25.0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from first dose of study treatment until the disease progression or death due to any cause per RECIST v.1.1 criteria. If date of progression or death occurred after more than 1 missed study visit, participants were censored at the time of last radiologic assessment prior to the missed visit. Participants without documented progression were also censored at the time of last radiologic assessment. Participants without any post baseline assessments were censored at date of start of study therapy.
Time Frame: From first dose of study treatment to time of disease progression or death, censored date (up to 23 months)
Population: Due to early termination, data for this outcome measure was not collected and analyzed.
Arm/Group | Arm 1: Selinexor
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants With Best Overall Response: RECIST v1.1 Criteria
Description: Best overall response rate was defined as the percentage of participants who achieved best response of CR, PR as assessed by the RECIST v1.1 criteria. CR was defined as disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taken as reference the baseline sum diameters.
Time Frame: From the date of first documented occurrence of response (CR or PR) until the date of documented progression or last disease assessment (up to 23 months)
Population: mITT population: Participants who received at least 1 dose of study drug and had at least 1 post-baseline efficacy assessment. In addition participants who received at least 1 dose of study drug, but discontinued treatment prior to first efficacy follow-up assessment due to death, toxicity, or disease progression were also included.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: Selinexor
Number analyzed (Participants) | 20
Percentage of participants | 0

4. Secondary Outcome: Absolute Values of Prostate Specific Antigen (PSA) Levels
Description: PSA marker was used for the assessment of disease progression and estimated the PSA level when compared to baseline.
Time Frame: Baseline, Day 1 of Cycles 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 (each cycle of 28 days) and End of Treatment (30 days after last dose of study treatment)
Population: mITT population was used for this outcome measure. Here, "number analyzed" signifies those participants who were evaluable for each specified time point.
Measure: Mean (Standard Deviation); unit: Microgram per liter (mcg/L)
Arm/Group | Arm 1: Selinexor
Number analyzed (Participants) | 20
Microgram per liter (mcg/L)
  Baseline | 253.54 (380.796)
  Cycle 2 Day 1: number analyzed (Participants) | 17
  Cycle 2 Day 1 | 1606.42 (5889.324)
  Cycle 3 Day 1: number analyzed (Participants) | 10
  Cycle 3 Day 1 | 204.64 (316.759)
  Cycle 4 Day 1: number analyzed (Participants) | 6
  Cycle 4 Day 1 | 160.50 (242.479)
  Cycle 5 Day 1: number analyzed (Participants) | 6
  Cycle 5 Day 1 | 199.70 (294.026)
  Cycle 6 Day 1: number analyzed (Participants) | 6
  Cycle 6 Day 1 | 253.95 (388.829)
  Cycle 7 Day 1: number analyzed (Participants) | 4
  Cycle 7 Day 1 | 264.40 (456.858)
  Cycle 8 Day 1: number analyzed (Participants) | 3
  Cycle 8 Day 1 | 417.93 (697.107)
  Cycle 9 Day 1: number analyzed (Participants) | 2
  Cycle 9 Day 1 | 17.90 (24.607)
  Cycle 10 Day 1: number analyzed (Participants) | 1
  Cycle 10 Day 1 | 1.30 (NA) — Standard deviation was not calculated due to single participant.
  Cycle 11 Day 1: number analyzed (Participants) | 1
  Cycle 11 Day 1 | 2.00 (NA) — Standard deviation was not calculated due to single participant.
  End of Treatment: number analyzed (Participants) | 14
  End of Treatment | 1026.43 (2155.744)

5. Secondary Outcome: Percent Change From Baseline in Prostate Specific Antigen Levels
Description: PSA marker was used for the assessment of disease progression and estimated the PSA level when compared to baseline.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change of PSA levels
Arm/Group | Arm 1: Selinexor
Number analyzed (Participants) | 20
percent change of PSA levels
  Cycle 2 Day 1: number analyzed (Participants) | 17
  Cycle 2 Day 1 | 210.74 (699.683)
  Cycle 3 Day 1: number analyzed (Participants) | 10
  Cycle 3 Day 1 | 80.31 (90.723)
  Cycle 4 Day 1: number analyzed (Participants) | 6
  Cycle 4 Day 1 | 30.51 (60.739)
  Cycle 5 Day 1: number analyzed (Participants) | 6
  Cycle 5 Day 1 | 187.86 (321.389)
  Cycle 6 Day 1: number analyzed (Participants) | 6
  Cycle 6 Day 1 | 281.05 (457.228)
  Cycle 7 Day 1: number analyzed (Participants) | 4
  Cycle 7 Day 1 | 327.46 (572.347)
  Cycle 8 Day 1: number analyzed (Participants) | 3
  Cycle 8 Day 1 | 92.37 (167.366)
  Cycle 9 Day 1: number analyzed (Participants) | 2
  Cycle 9 Day 1 | 1.43 (84.514)
  Cycle 10 Day 1: number analyzed (Participants) | 1
  Cycle 10 Day 1 | 8.33 (NA) — Standard deviation was not calculated due to single participant.
  Cycle 11 Day 1: number analyzed (Participants) | 1
  Cycle 11 Day 1 | 66.67 (NA) — Standard deviation was not calculated due to single participant.
  End of Treatment: number analyzed (Participants) | 14
  End of Treatment | 226.11 (200.131)

6. Secondary Outcome: Prostate Specific Antigen Response Rate
Description: PSA response rate was defined as number of participants who achieved a ≥30% drop in PSA at 12 Weeks when compared to baseline.
Time Frame: Baseline up to 12 weeks
Population: Analysis population included all participants from mITT population who had PSA data at 12 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Selinexor
Number analyzed (Participants) | 5
Participants | 1

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first dose of study treatment until death due to any cause. Participants who were still alive prior to the data cutoff for final efficacy analysis, or who dropout prior to study end, were censored at the day they were last known to be alive.
Time Frame: From first dose of study treatment to death, censored date (up to 23 months)
Population: Due to early termination, data for this outcome measure was not collected and analyzed.
Arm/Group | Arm 1: Selinexor
Number analyzed (Participants) | 0

8. Secondary Outcome: Pain Intensity Index (PPII) Total Score
Description: Quality of life (QoL) was assessed by verbal rating of participant's pain according to present pain intensity index. Participants were asked to describe "how severe their pain was at very moment". Present pain intensity was assessed on 5-point visual analog scale ranging from 0 to 5, where 0-no pain, 1-mild pain, 2-discomforting pain, 3-distressing pain, 4-horrible pain, and 5-excruciating pain. The higher scores indicated higher pain.
Time Frame: Baseline up to 30 days after last dose of study treatment (up to 23 months)
Population: Due to early termination, data for this outcome measure was not collected and analyzed.
Arm/Group | Arm 1: Selinexor
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) and Treatment Emergent Serious Adverse Events (TESAE)
Description: An adverse event (AE) was defined as the appearance of (or worsening of any pre-existing) undesirable sign, symptom, or medical condition that occur after participant's signed informed consent obtained. A serious adverse event (SAE) was defined as any AE, occurring at any dose (including after the informed consent form was signed and prior to dosing) that and regardless of causality that: results in death, is life-threatening (participant was at immediate risk of death from event as it occurred), requires in-patient hospitalization (formal admission to a hospital for medical reasons) or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect. TEAE was defined as any AE with onset or worsening of a pre-existing condition on or after the first administration of study treatment through 28 days following last dose or any event considered drug-related by the investigator through the end of the study.
Time Frame: From screening up to 23 months
Population: Safety population: All participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Selinexor
Number analyzed (Participants) | 20
Participants
  At least one TEAE | 20
  At least one TESAE | 9

ADVERSE EVENTS:
Time Frame: From screening up to 23 months
Description: Safety population consisted of all participants who received any amount of study drug.
Arm/Group | Arm 1: Selinexor
All-Cause Mortality (participants affected / at risk) | 10/20
Serious Adverse Events (participants affected / at risk) | 9/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Selinexor (N=20)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Influenza (Infections and infestations) | 1
Pneumonia Parainfluenzae Viral (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 2
Hemiparesis (Nervous system disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Selinexor (N=20)
Thrombocytopenia (Blood and lymphatic system disorders) | 16
Anaemia (Blood and lymphatic system disorders) | 12
Leukopenia (Blood and lymphatic system disorders) | 11
Lymphopenia (Blood and lymphatic system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 10
Abnormal Loss Of Weight (Metabolism and nutrition disorders) | 7
Decreased Appetite (Metabolism and nutrition disorders) | 7
Hyponatraemia (Metabolism and nutrition disorders) | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 5
Hypercreatininaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hyperamylasaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperlipasaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Anal Incontinence (Gastrointestinal disorders) | 2
Anal Paraesthesia (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 15
Oedema Peripheral (General disorders) | 3
Gait Disturbance (General disorders) | 1
Malaise (General disorders) | 1
Gamma-Glutamyltransferase Increased (Investigations) | 8
Aspartate Aminotransferase Increased (Investigations) | 7
Blood Alkaline Phosphatase Increased (Investigations) | 6
Alanine Aminotransferase Increased (Investigations) | 5
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 2
Hypersomnia (Nervous system disorders) | 2
Amnesia (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Insomnia (Psychiatric disorders) | 4
Confusional State (Psychiatric disorders) | 3
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Personality Change (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 7
Haemoglobinuria (Renal and urinary disorders) | 2
Nocturia (Renal and urinary disorders) | 2
Urinary Retention (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1
Hot Flush (Vascular disorders) | 2
Deep Vein Thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Venous Thrombosis (Vascular disorders) | 1
Vision Blurred (Eye disorders) | 3
Cataract (Eye disorders) | 1
Dry Eye (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Sinusitis (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Adrenal Insufficiency (Endocrine disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
This study was terminated due to enrollment challenges. The termination was not a consequence of any safety concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes